CLINICAL TRIAL: NCT03674476
Title: A Phase 1, Open-Label, Parallel-Group, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-986036 in Participants With Varying Degrees of Renal Function
Brief Title: An Investigational Study to Evaluate Experimental Medication BMS-986036 in Participants With Different Levels of Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB130-065; 2018-001497-19 (EudraCT Number)
Record Dates: First submitted 2018-08-29; First posted 2018-09-17 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: NAFLD; Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Pegbelfermin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Mild Renal Impairment (Experimental): The renal function will be defined by estimated glomerular filtration rate (eGFR) at Screening.
  Interventions: Drug: BMS-986036
- Moderate Renal Impairment (Experimental): The renal function will be defined by estimated glomerular filtration rate (eGFR) at Screening.
  Interventions: Drug: BMS-986036
- Severe Renal Impairment (Experimental): The renal function will be defined by estimated glomerular filtration rate (eGFR) at Screening.
  Interventions: Drug: BMS-986036
- Normal (Other): The renal function will be defined by estimated glomerular filtration rate (eGFR) at Screening.
  Interventions: Drug: BMS-986036

INTERVENTIONS:
Drug: BMS-986036 — Specified dose on specified days

SUMMARY:
This is an investigational study to evaluate the experimental medication BMS-986036 in participants with different levels of kidney function.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* BMI ≥ 25 and ≤ 40 kg/m2

Exclusion Criteria:

* Presence of any factors that would predispose the participant to infection (eg, extensive periodontal disease that warrants surgical or medical treatment, unhealed open wounds)
* Any bone trauma (fracture) or bone surgery (ie, hardware placement, joint replacement, bone grafting, or amputation) within 3 months of study drug administration
* Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status
* Any major surgery (eg, abdominal, thoracal, or cranial procedures) within 6 weeks of study drug administration
* Donation of blood or plasma to a blood bank, or in a clinical study (except at the screening visit) within 6 weeks of study drug administration
* Inability to tolerate subcutaneous injections

Other protocol defined inclusion/exclusion criteria could apply

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) of C-terminal intact BMS-986036 | Up to 30 days
Time of maximum observed serum concentration (Tmax) of C-terminal intact BMS-986036 | Up to 30 days
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of C-terminal intact BMS-986036 | Up to 30 days
Area under the serum concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of C-terminal intact BMS-986036 | Up to 30 days
Terminal elimination half-life (T-half) of C-terminal intact BMS-986036 | Up to 30 days
Apparent total body clearance (CLT/F) of C-terminal intact BMS-986036 | Up to 30 days
Apparent volume of distribution (Vz/F) of C-terminal intact BMS-986036 | Up to 30 days
Total renal clearance (CLR) of C-terminal intact BMS-986036 | Up to 30 days
Amount per fraction excreted into urine (Fe) of C-terminal intact BMS-986036 | Up to 30 days
Total amount excreted into urine (Ae) of C-terminal intact BMS-986036 | Up to 30 days

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of total BMS-986036 | Up to 30 days
Time of maximum observed serum concentration (Tmax) of total BMS-986036 | Up to 30 days
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of total BMS-986036 | Up to 30 days
Area under the serum concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of total BMS-986036 | Up to 30 days
Terminal elimination half-life (T-half) of total BMS-986036 | Up to 30 days
Apparent total body clearance (CLT/F) of total BMS-986036 | Up to 30 days
Apparent volume of distribution (Vz/F) of total BMS-986036 | Up to 30 days
Total renal clearance (CLR) of total BMS-986036 | Up to 30 days
Amount per fraction excreted into urine (Fe) of total BMS-986036 | Up to 30 days
Total amount excreted into urine (Ae) of total BMS-986036 | Up to 30 days
Incidence of injection site reactions (prospective) | Up to 30 days
Incidence of adverse events (AE) | Up to 30 days
Incidence of serious adverse events (SAE) | Up to 30 days
Incidence of clinically significant changes to events of special interest | Up to 30 days
  Events of special interest include injection site assessment, AEs leading to discontinuation, and deaths as well as AEs related to marked abnormalities in clinical laboratory tests, vital sign measurements, electrocardiogram (ECGs), and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Pharmaceutical Research Associates CZ, s.r.o, Prague, Czechia
- Hungary (3):
  - PRA Magyarorszag Kft, Budapest
  - Semmelweis Egyetem, Budapest
  - Clinical Research Unit Hungary, Miskolc

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm